CLINICAL TRIAL: NCT01942512
Title: Evaluation of Risk Factors Associated With Intracranial Aneurysm Recanalization After Endovascular Treatment
Brief Title: Risk Factors for Intracranial Aneurysm Recanalization After Endovascular Treatment.
Acronym: ARETA
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PN12145
Record Dates: First submitted 2013-09-11; First posted 2013-09-16 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Intracranial Aneurysm
Keywords: Intracranial Aneurysm - Endovascular treatment -; Coiling - Stenting - Flow diversion - Flow disruption -; Recanalization - Risk factors
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ARETA: All patients with intracranial aneurysms, ruptured or unruptured, treated by endovascular treatment
  Interventions: Device: Endovascular treatment of intracranial aneurysm

INTERVENTIONS:
Device: Endovascular treatment of intracranial aneurysm

SUMMARY:
Endovascular treatment is now the first line treatment for the management of intracranial aneurysms. However aneurysm recanalization is an important limitation to this treatment. Several factors seems to be associated with aneurysm recanalization including medical history of the patient, aneurysm status (ruptured or unruptured), aneurysm size and location, modalities of treatment, immediate post-operative occlusion of the aneurysm.

A precise knowledge of factors increasing the risk of aneurysm recanalization is quite important to optimize strategy of treatment and reduce the recanalization rate. No large, prospective, multicenter trial dealing with this question has been published in the literature.

DETAILED DESCRIPTION:
The prevalence of intracranial aneurysms is high (between 2 and 3%). The major risk of an intracranial aneurysm is its rupture leading to intracranial bleeding (subarachnoid, parenchymal and/or intraventricular) associated with mortality and morbidity.

Endovascular treatment is now the first line treatment for both ruptured and unruptured aneurysms. One major limitation of this treatment is aneurysm recanalization observed in approximately 20% of aneurysms and leading to retreatment in approximately 10% of aneurysms.

CARAT trial has shown that the risk of rebleeding after aneurysm coiling is significantly associated with the quality of aneurysm occlusion. The risk of rebleeding is 1.1% in case of complete occlusion, 2.9% when aneurysm occlusion is between 91 and 99%, 5.9% when aneurysm occlusion is between 70 et 90%, and 17.6% when aneurysm occlusion is less than 70%. However it should be outlined that few studies have clearly analyzed the relation between recanalization and rebleeding.

Several factors are probably associated with aneurysm recanalization. Ruptured aneurysms are more prone to aneurysm recanalization than unruptured aneurysm. Age, elevated blood pressure, smoking probably play a role in aneurysm recanalization. Anatomical features are also probably key factors for aneurysm recanalization. Aneurysm and neck sizes are probably important factors for aneurysm recanalization. The role of aneurysm location is more controversial. Therapeutic factors certainly play also an important role, but precise analyses are still missing. The quality of post-operative aneurysm occlusion is probably important for the future evolution of the aneurysm. Surface-modified coils have not demonstrated any efficacy to prevent aneurysm recanalization. The role of adjunctive techniques has also not precisely be evaluated (remodeling, stenting).

ELIGIBILITY:
Inclusion Criteria:

* Patients treated by endovascular approach for intracranial aneurysm(s)
* Patients older than 18 years
* Patients accepting to participate to the study

Exclusion Criteria:

* Patients younger than 18 years
* Patients protected by law
* Patients already treated by endovascular approach for an intracranial aneurysm
* Patients having a brain arteriovenous malformation
* Patients having a fusiform aneurysm
* Patients having a dissecting aneurysm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with intracranial aneurysms, ruptured or unruptured, treated by endovascular treatment
Sampling Method: Non-Probability Sample
Enrollment: 1275 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2017-06-23 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
aneurysm recanalization | assessed at 12 months

CONTACTS AND LOCATIONS:
Locations (22):
- France (22):
  - Centre Hospitalier Universitaire de Besançon, Besançon
  - CHU de Bordeaux, Bordeaux
  - CHU de CAEN, Caen
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - AP-HP, Hôpital Beaujon, Clichy
  - AP-HP, Hôpital Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - CHRU de LILLE, Lille
  - Hospices Civils de Lyon, Lyon
  - CHU de MONTPELLIER, Montpellier
  - CHU de Nancy, Nancy
  - CHU de Nantes, Nantes
  - CHU de Nice, Nice
  - Centre Hospitalier Sainte-Anne, Paris
  - AP-HP (Hôpital Pitié Salpétrière), Paris
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Centre Hospitalier Universitaire de Reims, Reims
  - CHU de Rennes, Rennes
  - CHU de Saint-Etienne, Saint-Etienne
  - Hopital Foch, Suresnes
  - CHU de Toulouse, Toulouse
  - CHU de Tours, Tours

REFERENCES:
- [Derived] Pierot L, Barbe C, Thierry A, Bala F, Eugene F, Cognard C, Herbreteau D, Velasco S, Chabert E, Desal H, Aggour M, Rodriguez-Regent C, Gallas S, Sedat J, Marnat G, Sourour N, Consoli A, Papagiannaki C, Spelle L, White P. Patient and aneurysm factors associated with aneurysm recanalization after coiling. J Neurointerv Surg. 2022 Nov;14(11):1096-1101. doi: 10.1136/neurintsurg-2021-017972. Epub 2021 Nov 5. PMID 34740986
- [Derived] Pierot L, Barbe C, Herbreteau D, Gauvrit JY, Januel AC, Bala F, Ricolfi F, Desal H, Velasco S, Aggour M, Chabert E, Sedat J, Trystram D, Marnat G, Gallas S, Rodesch G, Clarencon F, Papagiannaki C, White P, Spelle L; From the Departments of Neuroradiology, Research, and Public Health. Immediate post-operative aneurysm occlusion after endovascular treatment of intracranial aneurysms with coiling or balloon-assisted coiling in a prospective multicenter cohort of 1189 patients: Analysis of Recanalization after Endovascular Treatment of intracranial Aneurysm (ARETA) Study. J Neurointerv Surg. 2021 Oct;13(10):918-923. doi: 10.1136/neurintsurg-2020-017012. Epub 2020 Dec 21. PMID 33443137
- [Derived] Pierot L, Barbe C, Herbreteau D, Gauvrit JY, Januel AC, Bala F, Ricolfi F, Desal H, Velasco S, Aggour M, Chabert E, Sedat J, Trystram D, Marnat G, Gallas S, Rodesch G, Clarencon F, Papagiannaki C, White P, Spelle L. Delayed thromboembolic events after coiling of unruptured intracranial aneurysms in a prospective cohort of 335 patients. J Neurointerv Surg. 2021 Jun;13(6):534-540. doi: 10.1136/neurintsurg-2020-016654. Epub 2020 Sep 7. PMID 32895321
- [Derived] Pierot L, Barbe C, Herbreteau D, Gauvrit JY, Januel AC, Bala F, Ricolfi F, Desal H, Velasco S, Aggour M, Chabert E, Sedat J, Trystram D, Marnat G, Gallas S, Rodesch G, Clarencon F, Papagiannaki C, White P, Spelle L. Rebleeding and bleeding in the year following intracranial aneurysm coiling: analysis of a large prospective multicenter cohort of 1140 patients-Analysis of Recanalization after Endovascular Treatment of Intracranial Aneurysm (ARETA) Study. J Neurointerv Surg. 2020 Dec;12(12):1219-1225. doi: 10.1136/neurintsurg-2020-015971. Epub 2020 Jun 16. PMID 32546636
- [Derived] Pierot L, Barbe C, Ferre JC, Cognard C, Soize S, White P, Spelle L. Patient and aneurysm factors associated with aneurysm rupture in the population of the ARETA study. J Neuroradiol. 2020 Jun;47(4):292-300. doi: 10.1016/j.neurad.2019.07.007. Epub 2019 Sep 17. PMID 31539582